CLINICAL TRIAL: NCT06481670
Title: The Effects of Pre-operative Carbohydrate Fluids on PONV Incidence and Intensity in Orthognathic Surgery Patients
Brief Title: Carbohydrate Fluids and Post Operative Nausea and Vomiting
Acronym: PONV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-45096
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Nausea, Postoperative; Vomiting, Postoperative
Keywords: Orthognathic surgery; Carbohydrate rich drinks; Enhanced recovery after surgery (ERAS)
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative carbohydrate drink (Experimental): Participants randomized into this group will receive a carbohydrate drink before surgery.
  Interventions: Other: Carbohydrate drink
- Preoperative fasting (No Intervention): Participants randomized into this group will be fasting/nothing by mouth (NPO) before surgery.

INTERVENTIONS:
Other: Carbohydrate drink — The >50 g carbohydrate drink will be consumed up to 2 hours prior to surgery.
  Other Names: Apple juice
  Arms: Preoperative carbohydrate drink

SUMMARY:
This study is a prospective randomized clinical controlled trial testing the effects of pre-operative >50 g pre-operative carbohydrate fluids (apple juice) on a patient's post-operative nausea and vomiting (PONV) incidence and intensity. Optimizing fluid therapy in the peri-operative setting has been proven to improve patient outcomes and reduce complications and length of hospital stay. Based on practice guidelines under the American Society of Anesthesiologists, pre-operative hydration with complex carbohydrate drinks is safe and should be encouraged as it helps with improving metabolism to an anabolic state, decreases insulin resistance, reduces anxiety, and reduces PONV. While pre-operative carbohydrate (CHO) fluids have already been studied and adopted by other surgical specialities (Vascular, General Surgery, Orthopaedics, etc.), this has not yet been studied in oral and maxillofacial surgery, especially at Boston Medical Center (BMC).

During surgery, each participant will undergo our current Enhanced Recovery After Surgery "ERAS" protocol, which includes general anesthesia using inhalational gas, judicious IV fluids, intra-operative steroid and ondansetron (anti-emetic), use of 0.5% bupivacaine local anesthesia per quadrant at surgery end time, use of a throat pack, and orogastric/nasogastric (OG/NG) tube suctioning prior to extubation to minimize ingestion of blood. Pain and anxiety medications prior to and during surgery include 2 mg midazolam, fentanyl per anesthesia, toradol, and dexmedetomidine. Having this protocol will help minimize confounding variables that could affect the primary outcome-- incidence and severity of PONV.

The objectives for this research are:

* To evaluate if pre-operative clear CHO help reduce incidence and intensity of PONV.
* To assess if pre-operative clear carbohydrate fluids affect length of hospital stay
* To determine if pre-operative CHO reduce patient's pre-/post-operative anxiety
* To compare the amount/number of opioids and anti-emetics needed post-operatively between the two groups
* To compare ability for patients to return to PO hydration via the amount of fluid ingestion (mL) vs. if they need IV fluids due to decreased PO intake/inability to tolerate PO fluids
* To evaluate if patient Apfel score is also a strong indicator for incidence/severity of PONV

ELIGIBILITY:
Inclusion Criteria:

* Healthy, American Society of Anesthesiologists (ASA) I-II patients undergoing orthognathic surgery (single jaw, double jaw +/- adjunctive procedures including segmental Le Forts/genioplasty/septoplasty/turbinectomy)
* Operating room (OR) time scheduled prior to 12 pm

Exclusion Criteria:

* Non-English speaking/poor English comprehension
* Patient refusal
* Surgically Assisted Rapid Palatal Expansion (SARPE)
* Orthognathic surgery patients in addition to adjunctive procedures such as temporomandibular joint (TMJ) replacement, fat grafting, liposuction, or septorhinoplasty
* General Anesthesia using total IV anesthesia (TIVA)
* History of gastroesophageal reflux disease (GERD) or patient's with conditions that impair gastrointestinal (GI) motility
* History of motion sickness or postoperative nausea and vomiting (PONV)
* Hx of Diabetes Mellitus, endocrine disorders, or allergy to medications of the study
* Pre-operative scopolamine patch

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intensity of post operative nausea and vomiting (PONV) | 6 hours and 24 hours after surgery
  The post operative nausea and vomiting (PONV) intensity scale will be used to assess this outcome. It has 3 questions about nausea and vomiting and a question about the duration of nausea. Scores of 50 or greater are considered clinically important.
PONV based on the visual analog scale | 6 hours and 24 hours after surgery
  A visual analog scale from 0-10 (0= No nausea, 10= Worst possible nausea/vomiting) competed by the participant after surgery.

SECONDARY OUTCOMES:
The amount of opioids used for post operative pain | Discharge from hospital usually 1-2 days
  The amount of Oxycodone/Dilaudid will be abstracted from the electronic medical record (EMR) and converted and measured in morphine equivalents (MEQ)
The aount of anti-emetics used for PONV | Discharge from hospital usually1-2 days
  The amount of anti-emetics will be abstracted from the EMR
Frequency of emesis events | Discharge from hospital usually 1-2 days
  The frequency of emesis will be abstracted from the EMR
Post-operative fluid intake by mouth/per os (PO) | Discharge from hospital usually 1-2 days
  Post operative po fluids will be assessed in mL, abstracted from the EMR
Need for intravenous (IV) fluids | Discharge from hospital usually 1-2 days
  The number of participants who needed IV fluids will be abstracted from the EMR
Length of hospital stay | Discharge from hospital usually1-2 days
  The length of hospital stay in days will be abstracted from the EMR

OTHER OUTCOMES:
Patient Apfel Score | 9 months
  The simplified Apfel-score Scoring system will be used to assess risk of PONV. Scores can range from 0 to 4 based on these risk factors- Gender. Male= 0. Female=1; Smoking status. Smoker=0, Nonsmoker. =1; History of motion sickness or PONV. No= 0, Yes=1; Use of postoperative opioids. No=0, Yes=1. LoweV. The incidence of PONV, with the presence of 0, 1, 2, 3, and 4 risk factors is approximately 10%, 20%, 40%, 60%, and 80%, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Angeline Nguyen, DMD, Principal Investigator — Boston Medical Center, Oral and Maxillofacial Surgery
Locations (1):
- Boston Medical Center, Oral and Maxillofacial Surgey, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No